CLINICAL TRIAL: NCT03244436
Title: Emergency Surgery Following Pediatric Cardiac Catheterization
Brief Title: Emergency Surgery Following Pediatric Catheterization
Status: Completed | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed Kareem, Dr., Cairo University
Other Study IDs: Surgery after catheterization
Record Dates: First submitted 2017-08-07; First posted 2017-08-09 (Actual); Last update posted 2017-08-09 (Actual); Status verified 2017-08

CONDITIONS: Anesthesia

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Surgery following catheterization — Emergency surgery following pediatric cardiac catheterization

SUMMARY:
We study the outcome and prequesties of emergency surgeries that were necessary following accidents in the pediatric cardiac catheterization lab

ELIGIBILITY:
Inclusion Criteria:

* patients presenting for diagnostic or therapeutic pediatric cardiac catheterization

Exclusion Criteria:

* none

Ages: 2 Months to 9 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: 190 pediatric patients presenting for either diagnostic or interventional cardiac catheterization
Sampling Method: Non-Probability Sample
Enrollment: 190 (Actual)
Dates: Start 2013-06-15 (Actual); Primary Completion 2015-06-15 (Actual); Study Completion 2015-06-15 (Actual)

PRIMARY OUTCOMES:
Discharge from ICU | A 2 years study

IPD SHARING:
Plan to Share IPD: Undecided